CLINICAL TRIAL: NCT06527859
Title: Correlation Between Different Doses of Levothyroxine Supplementation and Peripheral Blood Th17/Treg Balance in Pregnant Women With Normal-high TSH and Positive TPOAb in the First Half of Pregnancy
Brief Title: Correlation Between Levothyroxine and Blood Th17/Treg in Pregnant Women With Normal-high TSH and Positive TPOAb
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to insufficient funding, rendering it impossible to continue purchasing reagents for experiments
Sponsor: Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xin Tian, Resident Physician, Third Affiliated Hospital of Zhengzhou University
Other Study IDs: ThirdZhengzhouU
Record Dates: First submitted 2024-07-14; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related; Thyroid Stimulating; Hormone, C
Keywords: levothyroxine; thyroid stimulating hormone; thyroid peroxidase antibodies; immunity; Th17/Treg
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The samples collected have no extra retention after being processed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: healthy pregnancy women
- disease group: pregnant women with normal-high TSH and positive TPOAb in the first half of pregnancy
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Levothyroxin — The disease group were divided into two groups ,25ugLT4 (HA group, n=17) and 50ugLT4 (HB group, n=17) respectively.
  Groups: disease group

SUMMARY:
The purpose of this clinical trial is to understand the impact of different doses of levothyroxine on the immune inflammatory response in pregnant women with normal-high TSH and positive TPOAb in the first half of pregnancy. It aims to answer the main questions:

Are there differences in immune inflammation between normal pregnant women and those in the disease group? Can different doses of levothyroxine improve the Th17/Treg ratio and cytokine levels in the disease group? Researchers first compared the differences between normal pregnant women and those in the disease group, and then administered two different doses of levothyroxine to the disease group to observe whether different doses of levothyroxine can improve the immune inflammation in this group.

pregnant women in the disease group will: Take the same dose of levothyroxine (25/50ug) every day Return for a follow-up visit after 4 weeks of medication

DETAILED DESCRIPTION:
To explore the correlation between different doses of levothyroxine (LT4) supplementation and Th17/Treg and cytokines in pregnant women with normal-high thyroid stimulating hormone (TSH) and positive thyroid peroxidase antibody (TPOAb) in the first half of pregnancy. From June 2022 to October 2023, 34 pregnant women with high- normal TSH and positive TPOAb in our hospital were selected (disease group), and 30 healthy pregnant women (control group) were matched; the disease group was divided into HA group and HB group according to the administration of 25 ug LT4 and 50 ug LT4. Blood samples were collected from the control group and the disease group before and 4-8 weeks after intervention to detect thyroid function, cytokine and blood lipid levels, flow cytometry to determine the proportion of Th17 and Treg cells, and methane hydrogen blowing examination was performed in parallel; the serological differences between the groups and before and after intervention were compared, and correlation analysis was used to analyze thyroid function, blood lipids, cytokines, and Th17/Treg.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid function level meets the specific reference range established by the laboratory department of our hospital based on the "Guidelines for the prevention and management of thyroid diseases during pregnancy and perinatal period" : FT4: 12-22pmol/L; disease group: TPOAb>;34IU/mL, TSH: 2.5mIU/L-upper limit of reference range; control group: TPOAb≤34IU/mL, TSH<2.5mIU/L;
* All pregnant women are in the first half of pregnancy (gestational age≤20 weeks).

Exclusion Criteria:

* Combined with hypothyroidism, subclinical hypothyroidism, and hyperthyroidism;
* Assisted reproduction;
* Multiple pregnancy;
* Combined with other autoimmune diseases such as antiphospholipid syndrome and thrombophilia;
* Severe intestinal diseases or intestinal surgery history, or the use of probiotics, prebiotics and other drugs that affect intestinal flora;
* Obesity, pre-pregnancy hyperlipidemia;
* Adverse reactions to LT4

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population that meets the inclusion and exclusion criteria and is willing to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Th17/Treg | 4 weeks
  Ratio of Th17 to Treg percentages in peripheral blood.

SECONDARY OUTCOMES:
cytokines, inflammatory factor | 4 weeks
  Concentrations of IL-2, 4, 6, 10, TNF-α, and hsCRP in peripheral blood.

OTHER OUTCOMES:
lipids, Small intestinal bacterial overgrowth | 4 weeks
  Concentrations ofTC, TG, LDL, HDL, FFA, ApoA, and ApoB in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Tian, Principal Investigator — Third Affiliated Hospital of Zhengzhou University; Yanjie Ban, Principal Investigator — Third Affiliated Hospital of Zhengzhou University
Locations (1):
- The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasa M, Contreras-Jurado C. Thyroid hormones act as modulators of inflammation through their nuclear receptors. Front Endocrinol (Lausanne). 2022 Aug 8;13:937099. doi: 10.3389/fendo.2022.937099. eCollection 2022. PMID 36004343
- [Background] Michalopoulou G, Alevizaki M, Piperingos G, Mitsibounas D, Mantzos E, Adamopoulos P, Koutras DA. High serum cholesterol levels in persons with 'high-normal' TSH levels: should one extend the definition of subclinical hypothyroidism? Eur J Endocrinol. 1998 Feb;138(2):141-5. doi: 10.1530/eje.0.1380141. PMID 9506856
- [Background] Cayres LCF, de Salis LVV, Rodrigues GSP, Lengert AVH, Biondi APC, Sargentini LDB, Brisotti JL, Gomes E, de Oliveira GLV. Detection of Alterations in the Gut Microbiota and Intestinal Permeability in Patients With Hashimoto Thyroiditis. Front Immunol. 2021 Mar 5;12:579140. doi: 10.3389/fimmu.2021.579140. eCollection 2021. PMID 33746942
- [Background] Xue H, Yu X, Ma L, Song S, Li Y, Zhang L, Yang T, Liu H. The possible role of CD4(+)CD25(high)Foxp3(+)/CD4(+)IL-17A(+) cell imbalance in the autoimmunity of patients with Hashimoto thyroiditis. Endocrine. 2015 Dec;50(3):665-73. doi: 10.1007/s12020-015-0569-y. Epub 2015 Mar 13. PMID 25771887
- [Background] undefined
- [Background] Xue H, Yang Y, Zhang Y, Song S, Zhang L, Ma L, Yang T, Liu H. Macrophage migration inhibitory factor interacting with Th17 cells may be involved in the pathogenesis of autoimmune damage in Hashimoto's thyroiditis. Mediators Inflamm. 2015;2015:621072. doi: 10.1155/2015/621072. Epub 2015 Mar 15. PMID 25861163
- [Background] Lee SY, Pearce EN. Assessment and treatment of thyroid disorders in pregnancy and the postpartum period. Nat Rev Endocrinol. 2022 Mar;18(3):158-171. doi: 10.1038/s41574-021-00604-z. Epub 2022 Jan 4. PMID 34983968
- [Background] Yetkin DO, Dogantekin B. The Lipid Parameters and Lipoprotein(a) Excess in Hashimoto Thyroiditis. Int J Endocrinol. 2015;2015:952729. doi: 10.1155/2015/952729. Epub 2015 May 3. PMID 26064115
- [Background] Sinha RA, Singh BK, Yen PM. Direct effects of thyroid hormones on hepatic lipid metabolism. Nat Rev Endocrinol. 2018 May;14(5):259-269. doi: 10.1038/nrendo.2018.10. Epub 2018 Feb 23. PMID 29472712
- [Background] Kim HJ, Park SJ, Park HK, Byun DW, Suh K, Yoo MH. Thyroid autoimmunity and metabolic syndrome: a nationwide population-based study. Eur J Endocrinol. 2021 Oct 11;185(5):707-715. doi: 10.1530/EJE-21-0634. PMID 34519275
- [Background] Ru X, Yang M, Teng Y, Han Y, Hu Y, Wang J, Tao F, Huang K. Association of maternal thyroid peroxidase antibody during pregnancy with placental morphology and inflammatory and oxidative stress responses. Front Endocrinol (Lausanne). 2023 Sep 22;14:1182049. doi: 10.3389/fendo.2023.1182049. eCollection 2023. PMID 37810887
- [Background] Mahto M, Chakraborthy B, Gowda SH, Kaur H, Vishnoi G, Lali P. Are hsCRP Levels and LDL/HDL Ratio Better and Early Markers to Unmask Onset of Dyslipidemia and Inflammation in Asymptomatic Subclinical Hypothyroidism? Indian J Clin Biochem. 2012 Jul;27(3):284-9. doi: 10.1007/s12291-012-0206-y. Epub 2012 Apr 18. PMID 26405389
- [Background] Cao Y, Jin X, Sun Y, Wen W. Therapeutic effect of mesenchymal stem cell on Hashimoto's thyroiditis in a rat model by modulating Th17/Treg cell balance. Autoimmunity. 2020 Feb;53(1):35-45. doi: 10.1080/08916934.2019.1697689. Epub 2019 Dec 3. PMID 31793369
- [Background] Vaivode I, Zake T, Strele I, Upmale-Engela S, Gogins D, Gersone G, Skesters A, Dambrova M, Konrade I. Stress-Related Immune Response and Selenium Status in Autoimmune Thyroid Disease Patients. Int J Mol Sci. 2023 Jan 26;24(3):2440. doi: 10.3390/ijms24032440. PMID 36768762
- [Background] Mazzieri A, Montanucci P, Basta G, Calafiore R. The role behind the scenes of Tregs and Th17s in Hashimoto's thyroiditis: Toward a pivotal role of FOXP3 and BACH2. Front Immunol. 2022 Dec 12;13:1098243. doi: 10.3389/fimmu.2022.1098243. eCollection 2022. PMID 36578493
- [Background] Xu Y, Zhao Y, Xu X, Yan Q, Yang L. Serum lipid profile in relation to free thyroxine and the effect of levothyroxine treatment on lipids in patients with isolated hypothyroxinemia during pregnancy: a single-center retrospective study. Lipids Health Dis. 2022 Dec 19;21(1):142. doi: 10.1186/s12944-022-01744-5. PMID 36536397
- [Background] Yu M, Long Y, Wang Y, Zhang R, Tao L. Effect of levothyroxine on the pregnancy outcomes in recurrent pregnancy loss women with subclinical hypothyroidism and thyroperoxidase antibody positivity: a systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2023 Dec;36(2):2233039. doi: 10.1080/14767058.2023.2233039. PMID 37433649
- [Background] Fenneman AC, Bruinstroop E, Nieuwdorp M, van der Spek AH, Boelen A. A Comprehensive Review of Thyroid Hormone Metabolism in the Gut and Its Clinical Implications. Thyroid. 2023 Jan;33(1):32-44. doi: 10.1089/thy.2022.0491. Epub 2023 Jan 6. PMID 36322786

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT06527859/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT06527859/ICF_001.pdf